CLINICAL TRIAL: NCT05239481
Title: Design and Clinical Application of Colonoscopy Position Identification Sheet: a Prospective, Multicenter, Randomized Controlled Study
Brief Title: Design and Clinical Application of Colonoscopy Position Identification Sheet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Chief of gastroenterology, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CPIS-LC
Record Dates: First submitted 2021-12-30; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Disease of Lower Digestive Tract; Nurse-Patient Relations
Keywords: colonoscopy; body position identification; bed sheet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Before the examination, the nurse chose the appropriate colonoscopy position size sheet according to the patient's age and body size and spread it on the examination bed; instructed the patient to lie in the designated area according to the body size.Description: ① take off your shoes; ② follow the bed chart; ③ fade your pants to your knees.
  Interventions: Device: colonoscopy position identification sheet
- control (Placebo Comparator): Traditional disposable cleaning sheets were used during control colonoscopy.Before the examination, the nursing staff took a unified and simple language to guide the patient, the following: ① please remove the shoes; ② please sit on the end of the bed mattress; ③ please lie to the left side; ④ please put the head close to the pillow; ⑤ please fade the pants to the knee; ⑥ please put the knee close to the abdomen.
  Interventions: Device: Traditional disposable cleaning sheet

INTERVENTIONS:
Device: colonoscopy position identification sheet — According to the body position requirements of the left lying position during colonoscopy, the research group used ink to add the body position prompt sign on the disposable bed sheet .Through the position identification, patients can intuitively understand the position that should be used in the operation and the position that should be placed in each part of the body.
  Arms: intervention
Device: Traditional disposable cleaning sheet — Traditional disposable cleaning sheets were used during control colonoscopy.Before the examination, the nursing staff took a unified and simple language to guide the patient.
  Arms: control

SUMMARY:
Before colonoscopy, the nursing staff need to educate the patient with posture coordination.However, it is difficult for some patients to understand the placement of the correct body position, which takes too much time to conduct repeated education, which wastes medical resources, reduces work efficiency, and even causes conflicts between doctors and patients.In this study, the colonoscopy position identification sheet with indicator function was designed to assist the position placement of patients. Preliminary experiments of small samples have achieved good clinical results. Now, multicenter, randomized controlled research is carried out to further verify the clinical application effect.

DETAILED DESCRIPTION:
This study was a prospective, multicenter, randomized controlled study involving patients who first underwent colonoscopy in 11 centers in China. Patients were randomly divided into two groups: the experimental group used colonoscopy position identification sheet, and the control group used ordinary clean sheets. The main evaluation index was the time required from the nurse guide to the patient complete the position placement, and the secondary indicators were doctors' satisfaction, nurse satisfaction and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 and signed informed consent
* with first colonoscopy
* with complete self-care (ADL 100)

Exclusion Criteria:

* patients with emergency colonoscopy
* communication or cognitive impairment
* patients requiring endoscopic intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
One-time success rate of body position placement | 30 minutes
  Refers to the proportion of the number of patients in the total study cases that can be accurately placed by the nurse
The time required for the nurse to guide it to complete the body position placement | 30 minutes
  The timing begins when the nurse began posture education, Until the patient correctly puts the required body position timing stops
Time for nurses to conduct physical position education | 30 minutes
  Refers to the length of the nurse to guide the completion of the body placement

SECONDARY OUTCOMES:
Satisfaction of doctors, nurses and patients | 5 minutes
  Scoring was performed using a visual simulation scale

REFERENCES:
- [Background] Zhao S, Yang X, Wang S, Meng Q, Wang R, Bo L, Chang X, Pan P, Xia T, Yang F, Yao J, Zheng J, Sheng J, Zhao X, Tang S, Wang Y, Wang Y, Gong A, Chen W, Shen J, Zhu X, Wang S, Yan C, Yang Y, Zhu Y, Ma RJ, Wang R, Ma Y, Li Z, Bai Y. Impact of 9-Minute Withdrawal Time on the Adenoma Detection Rate: A Multicenter Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e168-e181. doi: 10.1016/j.cgh.2020.11.019. Epub 2020 Nov 19. PMID 33220526